CLINICAL TRIAL: NCT02148965
Title: Effects of Exercise During Pregnancy on Maternal and Child Health: a Randomized Clinical Trial
Acronym: PAMELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, MARLOS RODRIGUES DOMINGUES, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAMELA-649.244; Wellcome Trust - 522.064 (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2014-05-22; First posted 2014-05-29 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Gestational Hypertension; Prematurity; Maternal Post-partum Depression; Maternal Post-partum Weight Retention; Child's Development
Keywords: motor activity; clinical trials; pregnancy; hypertension; cohort studies
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Premature Birth; Motor Activity; Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): Physical Exercise / Physical Activity. Exercise intervention, three weekly sessions. Each session will last around 60 minutes and will include aerobic exercises (treadmill or stationary cycling) and strength training (with focus on major muscle groups and pregnancy-specific exercises to help alleviate low back pain and work abdominal and pelvic floor muscles to prevent urinary incontinence).
  Interventions: Behavioral: Physical Exercise / Physical Activity
- Control Group (No Intervention): A group of eligible women, twice as large as the intervention group, will not receive the exercise intervention but will be followed-up equally to compare outcomes in the future.

INTERVENTIONS:
Behavioral: Physical Exercise / Physical Activity — Lifestyle intervention Exercise intervention, three weekly sessions. Each session will last around 60 minutes and will include aerobic exercises (treadmill or stationary cycling) and strength training (with focus on major muscle groups and pregnancy-specific exercises to help alleviate low back pain and work abdominal and pelvic floor muscles to prevent urinary incontinence).
  Arms: Lifestyle intervention

SUMMARY:
The Pamela Study is a clinical trial carried out during pregnancy to assess the potential effects of physical activity during pregnancy among previously inactive women. The trial is nested into a birth cohort of more than 4000 dyads (mother-child) and took place in Pelotas, Brazil.

DETAILED DESCRIPTION:
Introduction World Health Organization estimates that nearly 10% of births are preterm worldwide. In the city of Pelotas, based on previous population studies, the preterm birth rate is increasing (6.3% to 14.7% from 1982 to 2004). Preterm birth (PB) is a major public health issue as it is associated to most cases of neonatal deaths and its consequences are linked to later health outcomes.

One of the strongest predictors of PB is gestational hypertension (or eclampsia). PB risk and gestational hypertension may be altered by maternal behavior, such as leisure-time physical activity (LTPA), and overall maternal health influences the likelihood of both outcomes occurring. Biological plausibility lies on the fact that hypertension conditions are potentially influenced by LTPA directly or indirectly (as in the relation between excessive gestational weight gain and physical activity). Also, there is evidence that mental health plays a role in the determination of PB and, although biased by cross-sectional nature of studies, literature shows that physical activity may influence positively psychological aspects during pregnancy.

In Brazil less than 20% of pregnant women are physically active during leisure. Physical activity during pregnancy is associated to several characteristics resulting in improved health profiles that could potentially decrease hypertension occurrence and consequently preterm birth rates. However, few clinical trials have been carried out to study such relationship in representative population samples and many of the available evidence are based solely on observational studies.

Although early studies on the effects of leisure-time physical activity during pregnancy were concerned about potential harmful effects to the health of the mother and the fetus, these have not been proven over time. Currently, there is growing evidence supporting the safe promotion of physical activity during pregnancy targeting benefits to maternal and child health. However, most of the scientific evidence derives from observational studies. There is an urgent need for results from well-designed experimental studies that enable a better understanding of the impact of exercise during pregnancy on various health outcomes maternal and child.

Methodology The intervention will start after the 12th and before the 20th week of gestation and will last until the end of pregnancy or when women feel uncomfortable with the exercise routine. The intervention will consist of three weekly exercise sessions. Each session will last around 60 minutes and will include aerobic exercises (treadmill or stationary cycling) and strength training (with focus on major muscle groups and pregnancy-specific exercises to help alleviate low back pain and work abdominal and pelvic floor muscles to prevent urinary incontinence). Workouts will be guided and supervised by physical education professionals previously trained. The intensity of the exercises will be set according to woman's fitness level and will be altered according to the progress of pregnancy based on the perceived effort. All exercise sessions will take place at the School of Physical Education from the Federal University of Pelotas.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are at least in their 20th week of gestation, living in the city of Pelotas (Brazil), whose deliveries are due to 2015 and belonging to the 2015 Birth Cohort.

Exclusion Criteria:

* Hypertension
* Diabetes
* Preterm birth history
* Miscarriage history
* Heart disease
* In vitro fertilization
* Twin pregnancy
* Persistent bleeding
* Body mass index above 35kg/m2
* Heavy smokers (above 20 cigarettes/day)
* Active women (>150 min/week of physical activity).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Prematurity | Women will be interviewed at hospital soon after birth (up to 2 days after delivering)
  By the end of the intervention, after birth, the gestational age of each child will be measured to assess the preterm birth rate.

SECONDARY OUTCOMES:
Maternal post-partum depression | 3 months after the end of intervention
  A follow-up study will be carried out to assess post-partum maternal depression, comparing intervention and control women.
Child's development | Children will be followed-up and evaluated by the ages of 3, 12 and 24 months of age
  During the follow-up visits that will take place in the early years of childhood, children from mothers enrolled in the intervention/control groups will be compared with neurodevelopment screening tools.

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO C HALLAL, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Physical Education School, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Coll CVN, Domingues MR, Stein A, da Silva BGC, Bassani DG, Hartwig FP, da Silva ICM, da Silveira MF, da Silva SG, Bertoldi AD. Efficacy of Regular Exercise During Pregnancy on the Prevention of Postpartum Depression: The PAMELA Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186861. doi: 10.1001/jamanetworkopen.2018.6861. PMID 30646198
- [Derived] da Silva SG, Hallal PC, Domingues MR, Bertoldi AD, Silveira MFD, Bassani D, da Silva ICM, da Silva BGC, Coll CVN, Evenson K. A randomized controlled trial of exercise during pregnancy on maternal and neonatal outcomes: results from the PAMELA study. Int J Behav Nutr Phys Act. 2017 Dec 22;14(1):175. doi: 10.1186/s12966-017-0632-6. PMID 29273044
- [Derived] Domingues MR, Bassani DG, da Silva SG, Coll Cde V, da Silva BG, Hallal PC. Physical activity during pregnancy and maternal-child health (PAMELA): study protocol for a randomized controlled trial. Trials. 2015 May 24;16:227. doi: 10.1186/s13063-015-0749-3. PMID 26003406
- See also: Epidemiology Research Center — http://www.epidemio-ufpel.org.br